CLINICAL TRIAL: NCT06400082
Title: Investigating the Impact of Topical Insulin on Postoperative Wound Healing in Diabetic and Non-Diabetic Patients: A Randomized Controlled Trial
Brief Title: Topical Insulin for Postoperative Wound Healing
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omnia Azmy Nabeh, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-4-2023
Record Dates: First submitted 2024-04-26; First posted 2024-05-06 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Wound Complication; Insulin Resistance, Diabetes
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus | interventions — Insulin; Povidone-Iodine

STUDY DESIGN:
Intervention Model Description: 2 parallel groups, one treated with conventional povidone iodine 10% and the other is treated with topical insulin
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Povidone iodine 10% (Active Comparator)
  Interventions: Drug: Povidone-Iodine
- Topical insulin (Experimental)
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — Insulin is applied as a topical dressing for postoperative wounds and compared to the conventional povidone iodine treatment
  Arms: Topical insulin
Drug: Povidone-Iodine — Insulin is applied as a topical dressing for postoperative wounds and compared to the conventional povidone iodine treatment
  Arms: Povidone iodine 10%

SUMMARY:
This study aimed to investigate the potential effect of applying topical insulin therapy on the management and healing of postoperative wounds in patients known with type 2 diabetes mellitus (T2DM) and in a parallel group without diabetes. Investigators also studied the effect of topical insulin therapy on the expression of e-cadherin and Ki67, as markers for cellular proliferation and wound repair. The levels of IL-6 and the H2O2-induced DNA damage product, 8-hydroxy-2'-deoxyguanosine (8-OHdG), were assessed as markers for inflammation and oxidative stress. Finally, histomorphological assessment of skin biopsies was also carried out.

DETAILED DESCRIPTION:
The study participants will be recruited from general surgery department ,all patients with elective surgical procedure who will be admitted at the department for at least one week as it is the minimal duration of postoperative wound healing and the study will be conducted according to the regulations of ethical committee of clinical studies in the Faculty of Medicine, Cairo University

ELIGIBILITY:
Inclusion Criteria:

* Both males and females
* 40-60 years old
* diagnosed with type 2 DM (for the diabetic trial)
* For the diabetic trial: glycosylated hemoglobin (HBA1c) ≤7.5 %
* haemoglobin (Hb) ≥ 12 g/dl
* Patients who had a full thickness post-operative wound of ≥10 cm

Exclusion Criteria:

* Those with known history of immunodeficiency, keloid formation, or hyperkeratotic skin lesion.
* Patients who had hypersensitivity to insulin,
* Patients with severe infection,
* Patients with any severe organ dysfunction
* Patients who were admitted to ICU

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2023-04-16 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
Calculation of Unit Healing Time index | Before and after 7 days of therapy
  The total healing days and the surface area of the wound will be combined to report unit healing time in units

CONTACTS AND LOCATIONS:
Overall Officials: Omnia Azmy Nabeh, MD, Study Chair — Cairo University
Locations (1):
- Omnia Azmy Nabeh, Cairo, Egypt